CLINICAL TRIAL: NCT07306923
Title: Resilience Training Intervention: Its Effect on Parental Acceptance/Rejection and Burden of Children With Down Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24.03.250
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Down Syndrome
Keywords: resilience training; parental acceptance; parental burden; caregiver stress; behavioral intervention; psychological resilience; parental rejection
MeSH Terms: conditions — Down Syndrome; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Two-arm, non-randomized, parallel-group design comparing resilience training with usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience Training Intervention (experimental) (Experimental): Resilience Training Intervention
  Interventions: Behavioral: resilience training intervention
- Usual Care (Control) (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: resilience training intervention — A structured resilience training program delivered to parents of children with Down syndrome. The program consists of sessions designed to improve psychological resilience, enhance parental acceptance, and reduce caregiving burden. Training methods may include group discussions, skill-building exercises, and home practice tasks.
  Arms: Resilience Training Intervention (experimental)

SUMMARY:
This research will test whether a resilience training program can help parents of children with Down syndrome feel more accepting of their child and experience less caregiving burden.

Parents who care for a child with Down syndrome often face stress and emotional challenges. Building psychological resilience-the ability to adapt and recover from stress-may improve how parents cope and relate to their children.

The study will include about 50 parents of children with Down syndrome. Participants will be randomly assigned to one of two groups:

Experimental group: Receives the resilience training program.

Control group: Receives usual care.

Study phases

Before the program: Parents complete questionnaires that measure their resilience, their acceptance or rejection of their child, and their caregiving burden.

During the program: Parents in the experimental group attend a structured resilience training program based on their expressed needs.

After the program: The same questionnaires are repeated immediately after the program and again at a follow-up to see if any changes last.

The research hypothesis is that parents who take part in the resilience training will show higher acceptance, lower rejection, and reduced caregiving burden compared with parents who receive usual care.

This study will provide evidence on whether resilience training is a helpful, practical, and safe way to support families raising a child with Down syndrome.

DETAILED DESCRIPTION:
This quasi-experimental study will evaluate the effectiveness of a resilience training intervention on parental acceptance/rejection and caregiving burden among parents of children with Down syndrome.

Design

A non-randomized, controlled, pretest-posttest, repeated-measures design will be used. Approximately 50 parents will be allocated into an experimental group and a control group, based on availability and willingness to participate. Measurements will be taken at baseline, immediately post-intervention, and at follow-up.

Study Phases

Phase 1 - Needs assessment and program development

Assess baseline resilience, parental acceptance/rejection, and caregiving burden.

Develop and implement a tailored resilience training intervention based on identified needs.

Phase 2 - Evaluation

Evaluate the intervention's effect on parental acceptance/rejection.

Evaluate the intervention's effect on parental caregiving burden.

Intervention

The experimental group will receive a structured resilience training program designed to enhance coping skills, positive reframing, and stress management. The control group will continue with usual care during the same period.

Sample Size and Power

The required sample size was calculated a priori using G*Power 3.1.9.7 for a repeated-measures ANOVA (within-between interaction) with two groups and three time points.

Assuming a medium effect size (Cohen's f = 0.25), α = 0.05, power = 0.95, correlation among repeated measures = 0.50, and nonsphericity correction ε = 1.0, the analysis indicated 44 participants (22 per group).

To account for about 10% attrition, 50 participants (25 per group) will be recruited.

Expected Outcome

It is hypothesized that the resilience training will increase parental acceptance and reduce rejection and burden compared with usual care, despite the non-random allocation. Findings may guide family-centered mental-health programs for parents of children with Down syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Biological parent (mother or father) of a child (birth to 3 years old) diagnosed with Down syndrome.
* Age 18 years or older.
* Able to read and understand the study questionnaires and provide informed consent.
* Willing to attend all resilience training sessions (for the experimental group).
* parents who are not responsible for caring of any other patients in the family

Exclusion Criteria:

* Presence of severe mental illness (e.g., psychosis) or cognitive impairment that would hinder participation.
* Current enrollment in another structured psychological or parenting program aimed at resilience or acceptance.
* Any acute medical condition preventing attendance of the sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Parental Acceptance-Rejection scale | Baseline (pre-intervention), immediately post-intervention, and 1-month follow-up
  Mean change in parental acceptance-rejection score of parents of children with Down syndrome, measured using the Parental Acceptance-Rejection Questionnaire (PARQ) at baseline, immediately post-intervention, and 1-month follow-up.

SECONDARY OUTCOMES:
Change in Caregiver Burden Score | Baseline, immediately post-intervention, and 1-month follow-up
  Mean change in caregiver burden using Zarit Burden Interview at baseline, immediately post-intervention, and 1-month follow-up
Change in Maternal Resilience | Baseline, post-intervention, 1-month follow-up
  Mean change in maternal resilience measured using the Maternal Resilience Scale (MRS) at baseline, immediately post-intervention, and 1-month follow-up. Higher scores indicate greater resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Centre of Excellence which is affiliated to National Research Centre (NRC)., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided